CLINICAL TRIAL: NCT02345772
Title: Neoadjuvant Hormonal Therapy Combined With Chemoimmunotherapy (Taxotere, Trastuzumab and Pertuzumab) in Patients With HER2-positive and ER-Positive Breast Cancer (NeoHTTP Study)
Brief Title: Neoadjuvant Hormonal Therapy Combined With Chemoimmunotherapy
Acronym: Neohttp
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI no longer at site. Data was not collected
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB 20140462
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: HER2-positive Breast Cancer; ER-positive Breast Cancer
MeSH Terms: interventions — Fulvestrant; Docetaxel; Trastuzumab; Protons; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Protocol (Experimental): Hormonal therapy with fulvestrant 500 mg will be administered intramuscularly on days 1, 15 of the first cycle, and thereafter on day 1 of every 28-day cycle for up to 5 cycles before surgery. Docetaxel (T) 75 mg/m2 every 3 weeks will be given for four cycles. Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent cycles before and after surgery), pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery.
  Interventions: Drug: fulvestrant 500 mg; Drug: Docetaxel; Drug: Trastuzumab (H, 8mg/kg; Drug: Pertuzumab (P, 840 mg

INTERVENTIONS:
Drug: fulvestrant 500 mg — Hormonal therapy with fulvestrant 500 mg will be administered intramuscularly on days 1, 15 of the first cycle, and thereafter on day 1 of every 28-day cycle for up to 5 cycles before surgery.
  Other Names: fulvestrant
Drug: Docetaxel — Docetaxel (T) 75 mg/m2 every 3 weeks will be given for four cycles.
  Other Names: Taxotere
Drug: Trastuzumab (H, 8mg/kg — Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent cycles before and after surgery), pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery.
  Other Names: Trastuzumab
Drug: Pertuzumab (P, 840 mg — Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent cycles before and after surgery), pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery.
  Other Names: Pertuzumab

SUMMARY:
Hormonal therapy administered before surgery in ER-positive and HER2-positive patients with breast cancer.

DETAILED DESCRIPTION:
Hormonal therapy with fulvestrant 500 mg to be administered before surgery With docetaxel, Trastuzumab, and pertuzumab to determine pathological complete remission rate at the time of surgery in ER-positive and HER2-positive patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with histologically, and radiographically confirmed non-metastatic ER-positive (defined as ≥30% of positive cells) and HER2-positive (defined as overexpression by immunohistochemistry (3+) or 2+ and positive by defined by fluorescence or dual in situ hybridization.) breast cancer with minimal tumor size over 2 cm (≥T2 lesion) to receive neoadjuvant chemotherapy recommended by the treating physician
2. Eastern Cooperative Oncology Group (ECOG) performance status score < 1
3. Absolute neutrophil count > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 8.5 g/dL
4. Serum creatinine ≤1.5 times the upper limit of the normal range, total bilirubin ≤ 1.5 X ULN (≤ 3 mg/dL if clinically diagnosed with Gilbert syndrome) AST/ALT ≤ 2.5 X ULN (AST/ALT ≤ 5X ULN if clinically diagnosed with Gilbert syndrome)
5. Women of child-bearing potential (i.e., women who are pre-menoposaul or not surgically sterile) must have a negative serum pregnancy test within 2 weeks prior to beginning treatment

Exclusion Criteria:

1. Uncontrolled cardiac disease, such as angina, hypertension or significant arrhythmias
2. LVEF (left ventricular ejection fraction) < 50% on any prior assessment. Note: Assessment of LVEF is done before and after trastuzumab-based chemotherapy as standard of care
3. Pregnant or lactating females
4. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements
5. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, FNP, Study Director — Research Director
Locations (1):
- Western Regional Medical Center, Inc., Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Protocol: Hormonal therapy with fulvestrant 500 mg will be administered intramuscularly on days 1, 15 of the first cycle, and thereafter on day 1 of every 28-day cycle for up to 5 cycles before surgery. Docetaxel (T) 75 mg/m2 every 3 weeks will be given for four cycles. Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent cycles before and after surgery), pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery.
  fulvestrant 500 mg: Hormonal therapy with fulvestrant 500 mg will be administered intramuscularly on days 1, 15 of the first cycle, and thereafter on day 1 of every 28-day cycle for up to 5 cycles before surgery.
  Docetaxel (T) 75 mg/m2 (Taxotere): Docetaxel (T) 75 mg/m2 every 3 weeks will be given for four cycles.
  Trastuzumab (H, 8mg/kg: Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent cycles before and after surgery), pertuzumab (P, 840 mg for 1st cycle,
Period: Overall Study
Arm/Group | Treatment Protocol
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected. No study data was collected
Arm/Group | Treatment Protocol
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Remission Rate
Description: To determine pathological complete remission rate at the time of surgery in ER-positive and HER2-positive breast cancer patients undergoing neoadjuvant chemoimmunotherapy (docetaxel, trastuzumab, pertuzumab) concurrently with neoadjuvant hormonal therapy with fulvestrant. Note: pCR, defined as the absence of invasive neoplastic cells of the primary tumor in the breast, remaining in-situ lesions are allowed, ypT0-is;
Time Frame: one year
Population: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Arm/Group | Treatment Protocol
Number analyzed (Participants) | 0

2. Secondary Outcome: Partial Pathological Response Rate
Description: Partial pathological response rate at the time of surgery and biomarker changes in breast cancer (biopsy vs residual tumor) before and after neoadjuvant chemotherapy Note: pPR, defined as residual invasive disease of 1cm, ypT1a-b.
Time Frame: One Year
Population: as for outcome 1
Arm/Group | Treatment Protocol
Number analyzed (Participants) | 0

3. Secondary Outcome: QTA (Quantitative Texture Analysis)
Description: QTA (Quantitative Texture Analysis): will be obtained from baseline mammogram and the correlation with clinical outcome after neoadjuvant therapy will be performed.
Time Frame: One year
Population: as for outcome 1
Arm/Group | Treatment Protocol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Description: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Arm/Group | Treatment Protocol
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes